CLINICAL TRIAL: NCT06466044
Title: Effect and Mechanism of Auricular Acupressure on Insomnia in Patients With Functional Dyspepsia：a Randomized Clinical Trial
Brief Title: Effect and Mechanism of Auricular Acupressure on Functional Dyspepsia With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-KLS-231-05
Record Dates: First submitted 2024-05-14; First posted 2024-06-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Functional Dyspepsia; Insomnia
Keywords: Auricular Acupressure; Functional Dyspepsia; insomnia; clinical efficacy; Effect mechanism study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: the two groups affixed the auricular points with Vaccaria seed to the ear, the control group affixed to the ear lobe, and the experimental group affixed to the ear nail area. The ear compression treatment was performed, and the pressure was subject to the patient's gas state (acid, numbness, weight, swelling, etc.). Frequency: 3 times a day, press the ear point within half an hour after a meal, the press frequency is about 30 times, and the bilateral ear lobe is alternately pressed. The treatment lasted for 2 weeks. Go to the hospital once a week to change the ear patch.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During clinical trials, subjects, evaluators, data managers, and statisticians are unaware of treatment assignments. After randomization and allocation by an independent data manager, it is handed over to the nurse, who will not be involved in the results evaluation or data analysis. Neither the study participants nor the investigators had any effect on randomization and assigned hiding. The participants were told there were two treatment options. Two months after the study, patients were asked to complete a blind assessment and a perceived efficacy assessment, and were asked to guess which treatment they had received to test the success of the blind. All researchers will receive training on the methodological specifications of this study prior to the trial and strictly adhere to the principle of task separation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Auricular point containing Vaccaria seed was attached to the auricular concha area rich in vagus nerve. Frequency: Press the auricular points three times a day within half an hour after meals, and press the auricular points for about 30 times. Press the auricular concha alternately. The treatment lasted for 2 weeks. Go to the hospital once a week to change the ear patch.
  Interventions: Behavioral: Auricular acupressure in concha area
- Control group (Sham Comparator): Auricular point with Vaccaria seed was attached to the earlobe, which is the place with the least vagal innervation. Frequency: Press the auricular points three times a day within half an hour after meals, and press the auricular points for about 30 times. Press the bilateral earlobes alternately. The treatment lasted for 2 weeks. Go to the hospital to change the ear patch once a week.
  Interventions: Behavioral: Auricular acupressure in earlobe

INTERVENTIONS:
Behavioral: Auricular acupressure in concha area — The method of pressing beans on auricular points is based on the meridian theory and viscera theory in the basic theory of traditional Chinese medicine, combined with the knowledge of modern medical anatomy, and from the perspective of syndrome differentiation and treatment, relevant auricular points are selected, and appropriate stimulation such as kneading, pressing, pinching and pressing is given to the seeds of Vaccaria seed attached to the concha auricularis, so that the auricular points can produce acid, numbness, swelling and pain slowly and continuously. For therapeutic purposes.
  Arms: Treatment group
Behavioral: Auricular acupressure in earlobe — The auricular point pressing bean method is based on the meridian theory and viscera theory in the basic theory of traditional Chinese medicine, combined with the knowledge of modern medical anatomy, and from the perspective of syndrome differentiation and treatment, the relevant auricular points are selected, and the seeds attached to the ear lobe, which is the least innervated part of vagus nerve, are given appropriate stimulation such as kneading, pressing, pinching and pressing, so that the auricular points produce acid, numbness, swelling and pain slowly and continuously. For therapeutic purposes.
  Arms: Control group

SUMMARY:
Functional dyspepsia refers to a chronic digestive system disease with upper abdominal symptoms originating from the gastroduodenal region, and after clinical examination, including upper gastrointestinal endoscopy, the organic diseases causing the above symptoms are excluded. According to Rome IV standard, functional dyspepsia can be divided into two categories: postprandial discomfort syndrome and epigastric pain syndrome. FD not only seriously affects the quality of life of patients, but also causes a heavy social and economic burden. Therefore, active prevention and treatment of FD, especially PDS, has become an unavoidable problem in clinic.

Epidemiological investigation shows that about 30% FD patients have many negative emotions such as insomnia, anxiety and depression, and many anti-negative emotional drugs themselves can cause gastrointestinal side effects, which are considered to be the key reasons for the recurrence of symptoms. In recent years, people have paid more and more attention to the brain-gut axis. Microbial-intestinal-brain axis can also affect brain function by releasing neurotransmitters and inflammatory mediators. In addition, the interaction between bile acids and intestinal microflora may also affect the normal function of the intestine. However, the relationship between specific bile acids, microflora and functional dyspepsia is still uncertain.

At present, the effective and safe treatment methods for FD with insomnia are still very limited. In recent years, Auricular Acupressure has obvious advantages in treating FD with insomnia. This study plans to study the clinical efficacy and mechanism of Auricular Acupressure on functional dyspepsia with insomnia. Provide more treatment methods and ideas for clinicians, popularize and apply green diagnosis and treatment methods, bring good news to more patients, and produce remarkable economic and social benefits

DETAILED DESCRIPTION:
1. The effective rate. The effective rate was based on the proportion of patients whose PSQI score of ≥ 50% at 2 weeks as compared with the baseline
2. PSQI score. The PSQI is a widely used questionnaire to assess one's sleep quality for the past month, with 7 components for 7 specific features of sleep.
3. sleep quality assessed by actigraphy: Objectively record the clinical sleep changes of the patients before and after treatment by the ActiGraph wGT3X-BT.
4. modified FDSD
5. SF-NDI: Evaluate the functional dyspepsia of patients with functional dyspepsia and insomnia by SF-NDI.
6. SAS, SDS: SAS and SDS were used to evaluate the patients' psychological status.
7. HAS, HRV: Assess the autonomic nervous function of patients before and after treatment by the excessive arousal scale and heart rate variability.
8. To study the therapeutic mechanism of patients before and after treatment by detecting fecal intestinal microecological flora and Short-chain fatty acid spectrum metabonomics.
9. The changes of tongue and pulse before and after treatment were detected by tongue and pulse meter
10. Averse events. Any adverse events, such as unfavorable or unintended signs, symptoms, or diseases, related to the AA treatment or the administration of these comorbidity was reported by patients and professional nurses. Severe adverse events had to be reported to the principal investigator and the data and safety monitoring board within 24 hours after their occurrence.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of functional dyspepsia and insomnia
* Age 18 years or older
* The following drugs were not taken for at least 2 weeks before enrollment: antibiotics (oral, intramuscical and intravenous), microecological preparations (probiotics, prebiotics and Biostime, etc.) and other drugs affecting the gastrointestinal flora, any drugs or health products that improve sleep quality or inhibit neural activity in the brain, drugs related to the treatment of functional dyspepsia or other related treatments
* Agree to participate in the study voluntarily and sign the informed consent

Exclusion Criteria:

1. Secondary insomnia caused by medication or other diseases;
2. Patients with comorbid mental disorders, as well as severe diseases of the heart, liver, kidneys and other systems;
3. Those who have previously received this treatment method or participated in other clinical trials within 6 months;
4. Presence of contraindications for auricular patches, such as skin hypersensitivity or damage to the application site;
5. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
the effective rate at week 2 | 2-week
  The effective rate was based on the proportion of patients whose PSQI score of ≥ 50% at 2 weeks as compared with the baseline PSQI score

SECONDARY OUTCOMES:
the effective rate at week 8 | 8-week after treatment
  The effective rate was based on the proportion of patients whose PSQI score of ≥ 50% at 8 weeks as compared with the baseline PSQI score
short form-Nepean dyspepsia Index | baseline, 2 weeks, 8 weeks after treatment
  Clinical functional dyspepsia was assessed by the short form-Nepean dyspepsia Index scale. The short form-Nepean dyspepsia Index scale is scored using a 5-point Likert scale (1-5 points), with the lowest score of 10 points and the highest score of 50 points.
Pittsburgh Sleep Quality Index | baseline, 2 weeks, 8 weeks after treatment
  Clinical sleep was assessed by the Pittsburgh Sleep Quality Index. This scale is scored on a scale of 0-3, with a cumulative score of PQSI total score (0-21) and a maximum score of 21. The higher the score, the worse the quality of sleep.
Self-rated Anxiety Scale | baseline, 2 weeks, 8 weeks after treatment
  Clinical sleep was assessed by the Self-rated Anxiety Scal.The anxiety self-rating scale is scored on a 4-point scale, with a maximum score of 100 and a minimum score of 20. The higher the score, the more severe the anxiety symptoms. A score below 50 is normal; 50-60 is mild; A score of 70 or more is considered severe.
Self-rated Depression Scale | baseline, 2 weeks, 8 weeks after treatment
  Clinical sleep was assessed by the Self-rated Depression Scale. The depression self-rating scale is scored on a 4-point scale, with a maximum score of 100 and a minimum score of 20. The higher the score, the more severe the depressive symptoms. A score of 53-62 is mild depression, 63-72 is moderate depression, and a score above 72 is severe depression.
Hyperarousal scale | baseline, 2 weeks, 8 weeks after treatment
  Changes in autonomic nervous function before and after treatment were evaluated on Hyperarousal scale
Heart rate variability | baseline, 2 weeks, 8 weeks after treatment
  Changes in autonomic nervous function before and after treatment were evaluated on Hyperarousal scale
Sleep efficiency | baseline, 2 weeks, 8 weeks after treatment
  We will collect the sleep efficiency of patients before and after treatment by ActiGraph wGT3X-BT. >85% indicates good sleep quality. 85% or less indicates poor sleep quality.
Total sleep time. | baseline, 2 weeks, 8 weeks after treatment
  We will collect the total sleep time of patients before and after treatment by ActiGraph wGT3X-BT. An increase in total sleep time indicates improved sleep quality.
Wake After Sleep Onset | baseline, 2 weeks, 8 weeks after treatment
  We will collect the post-sleep awakening time of patients before and after treatment by ActiGraph wGT3X-BT. Increased waking after sleep onset suggests poorer sleep quality.
Sleep fragmentation index | baseline, 2 weeks, 8 weeks after treatment
  We will collect the sleep fragmentation index of patients before and after treatment by ActiGraph wGT3X-BT. An increase in the sleep fragmentation index indicates poor sleep quality.
OTE | baseline, 2 weeks, 8 weeks after treatment
  To assess patient satisfaction with treatment of functional dyspepsia
modified FDSD, | baseline, 2 weeks, 8 weeks after treatment
  The patient was evaluated for symptoms of functional dyspepsia

OTHER OUTCOMES:
Changes in the composition of the intestinal microbiota. | baseline,2 weeks after treatment, 8 weeks after treatment
  Stool samples were collected, and the changes of intestinal microbiota components before and after treatment were explored by analyzing the microbial composition, diversity index, and species composition of intestinal microbiota in feces
Changes in Short-chain fatty acid profile composition. | baseline,2 weeks after treatment, 8 weeks after treatment
  Blood samples were collected to analyze the changes in the quantity and concentration of short-chain fatty acids in blood, and to explore the changes in the composition of short-chain fatty acids spectrum before and after treatment
Adverse event table | baseline,2 weeks after treatment, 8 weeks after treatment
  Patient safety during treatment was assessed by the Adverse Events Table

CONTACTS AND LOCATIONS:
Overall Officials: Wu JianNong, doctor, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen MY, Li ZJ, Zhou R, Lou QY, Ying ZK, Liu S, Feng DD, Yang DD, Jiang LX, Wang XL, Wu JX, Li M, Wu JN. Efficacy and Safety of Auricular Acupressure for Insomnia in Patients With Functional Dyspepsia: A Randomized Controlled Trial. Am J Gastroenterol. 2025 Dec 10. doi: 10.14309/ajg.0000000000003880. Online ahead of print. PMID 41369283
- [Derived] Shen MY, Lou QY, Liu S, Li ZJ, Lin TC, Zhou R, Feng DD, Yang DD, Wu JN. The efficacy and safety of auricular acupoint therapy on treating functional dyspepsia with insomnia: study protocol for a randomized controlled trial. Front Med (Lausanne). 2025 Mar 12;12:1496502. doi: 10.3389/fmed.2025.1496502. eCollection 2025. PMID 40144883

DOCUMENTS (1):
  • Informed Consent Form (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT06466044/ICF_000.pdf